CLINICAL TRIAL: NCT01933334
Title: The LOTUSS Trial: An Open-Label, Randomized, Phase 2 Study of the Safety and Tolerability of Pirfenidone When Administered to Patients With Systemic Sclerosis-Related Interstitial Lung Disease (SSc-ILD) (LOTUSS)
Brief Title: Safety and Tolerability of Pirfenidone in Participants With Systemic Sclerosis-Related Interstitial Lung Disease (SSc-ILD) (LOTUSS)
Acronym: LOTUSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSSc-001
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Systemic Sclerosis
Keywords: pirfenidone; SSc-ILD; scleroderma; systemic sclerosis; interstitial lung disease
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pirfenidone: 4-Week Titration Group (Experimental): Participants will receive one 267 milligrams (mg) oral pirfenidone capsule three times daily (TID) (801 mg per day [mg/day]) for 2 weeks followed by two 267 mg oral pirfenidone capsules TID (1602 mg/day) for 2 weeks (titration period) and then three 267 mg oral pirfenidone capsules TID (2403 mg/day) for 12 weeks maintenance period).
  Interventions: Drug: Pirfenidone
- Pirfenidone: 2-Week Titration Group (Experimental): Participants will receive one 267 mg oral pirfenidone capsule TID (801 mg/day) for 1 week followed by two 267 mg oral pirfenidone capsules TID (1602 mg/day) for 1 week (titration period) and then three 267 mg oral pirfenidone capsules TID (2403 mg/day) for 14 weeks (maintenance period).
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be administered orally at a dose of 267 mg one oral capsule TID (801 mg/day) for 1 or 2 weeks followed by two 267 mg oral capsules TID (1602 mg/day) for 1 or 2 weeks (titration period) and then three 267 mg oral capsules TID (2403 mg/day) for 12 weeks (maintenance period).

SUMMARY:
PSSc-001 (LOTUSS)

This study is a Phase 2, multinational, open-label, randomized, parallel-group, safety and tolerability study of pirfenidone in participants with systemic sclerosis-related interstitial lung disease (SSc-ILD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of systemic sclerosis-related (SSc) confirmed by the American College of Rheumatology classification criteria of systemic sclerosis (Masi 1980); duration of diagnosis less than (<) 7 years
2. Diagnosis of SSc-ILD based on an high-resolution computed tomography (HRCT) scan
3. Screening forced vital capacity (FVC) greater than equal to (>=) 50 percent (%) of the predicted value, and screening carbon monoxide diffusing capacity (DLCO) >=40% of the predicted value
4. At study entry, the participant either was not taking SSc-ILD medication or was taking cyclophosphamide or mycophenolate

Exclusion Criteria:

1. Clinically significant pulmonary hypertension
2. Known underlying liver disease
3. Clinical evidence of significant aspiration or uncontrolled gastroesophageal reflux
4. History of clinically significant asthma or chronic obstructive pulmonary disease
5. Active infection
6. Diagnosis of another connective tissue disorder
7. Evidence of a malignancy that is likely to result in significant disability or require significant medical or surgical intervention
8. History of unstable or deteriorating cardiac or pulmonary disease (other than SSc-ILD)
9. Pregnancy or lactation
10. Creatinine clearance <40 milliliters per minute (mL/min)
11. Prior use of pirfenidone
12. Unsuitable for enrollment or unlikely to comply with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: For additional information, call InterMune Medical Information Telephone: 1-888-486-6411, Study Chair — University of Cincinnati
Locations (22):
- United States (18):
  - Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University School of Medicine, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Chicago, Illinois
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hospital for Special Surgery, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University South Carolina, Charleston, South Carolina
  - University of Texas, Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Italy (2):
  - Università di Torino, Orbassano, Turin
  - University of Florence, Florence

REFERENCES:
- [Background] Preliminary criteria for the classification of systemic sclerosis (scleroderma). Subcommittee for scleroderma criteria of the American Rheumatism Association Diagnostic and Therapeutic Criteria Committee. Arthritis Rheum. 1980 May;23(5):581-90. doi: 10.1002/art.1780230510. PMID 7378088
- [Derived] Khanna D, Albera C, Fischer A, Khalidi N, Raghu G, Chung L, Chen D, Schiopu E, Tagliaferri M, Seibold JR, Gorina E. An Open-label, Phase II Study of the Safety and Tolerability of Pirfenidone in Patients with Scleroderma-associated Interstitial Lung Disease: the LOTUSS Trial. J Rheumatol. 2016 Sep;43(9):1672-9. doi: 10.3899/jrheum.151322. Epub 2016 Jul 1. PMID 27370878

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone: 2-Week Titration Group: Participants received one 267 milligrams (mg) oral pirfenidone capsule three times daily (TID) (801 mg per day [mg/day]) for 1 week followed by two 267 mg oral pirfenidone capsules TID (1602 mg/day) for 1 week (titration period) and then three 267 mg oral pirfenidone capsules TID (2403 mg/day) for 14 weeks (maintenance period).
- Pirfenidone: 4-Week Titration Group: Participants received one 267 mg oral pirfenidone capsule TID (801 mg/day) for 2 weeks followed by two 267 mg oral pirfenidone capsules TID (1602 mg/day) for 2 weeks (titration period) and then three 267 mg oral pirfenidone capsules TID (2403 mg/day) for 12 weeks (maintenance period).
Period: Overall Study
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group
Started | 32 | 31
Completed | 27 | 29
Not Completed | 5 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who provided written informed consent and received at least one dose of study medication.
Groups:
- Pirfenidone: 2-Week Titration Group: Participants received one 267 mg oral pirfenidone capsule TID (801 mg/day) for 1 week followed by two 267 mg oral pirfenidone capsules TID (1602 mg/day) for 1 week (titration period) and then three 267 mg oral pirfenidone capsules TID (2403 mg/day) for 14 weeks (maintenance period).
- Total: Total of all reporting groups
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12.08) | 51.9 (12.52) | 50.6 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs)
Description: Percentage of participants who had treatment-emergent AEs, defined as newly occurring or worsening after first dose. Relatedness to (study drug) was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: From baseline up to 28 days after the last dose of study drug (last dose = Week 16)
Population: Safety population included all randomized participants who provided written informed consent and received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group
Number analyzed (Participants) | 32 | 31
percentage of participants | 96.9 | 96.8

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From baseline up to 28 days after the last dose of study drug (last dose = Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group
Number analyzed (Participants) | 32 | 31
percentage of participants | 9.4 | 0.0

3. Secondary Outcome: University of California at Los Angeles (UCLA) Scleroderma Clinical Trial Consortium (SCTC) Gastrointestinal Trial (GIT) Questionnaire Scale Scores
Description: UCLA SCTC GIT Scale 2.0 is a 34-item self-administered questionnaire to obtain participant's assessment of the frequency of GI symptoms in preceding 7 days and how symptoms affected his/her life. All but 2 items were scored on a 0 to 3 scale (0=better health, 3=worse health); remaining 2 items were scored as 0 (better health) and 1 (worse health). The 34 items are divided into seven scales (reflux, distention/bloating, fecal soilage, diarrhea, social functioning, emotional well-being, and constipation). Individual scale score was calculated as the average of the items in the scale. Individual scale score ranged from 0 to 3 for reflux, distention/bloating, fecal soilage, social functioning, and emotional well-being; 0 to 2 for diarrhea; and 0 to 2.5 for constipation. A total score was also calculated as the average of 6 of the 7 scales (omitting constipation) and ranged from 0 to 2.83. For individual and total scores 0 indicated better health and higher score indicates worse health.
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: Safety population. n = number of participants analyzed at specified time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group
Number analyzed (Participants) | 32 | 31
units on a scale
  Reflux: Baseline (n=32, 31) | 0.3398 (0.34083) | 0.3347 (0.29117)
  Reflux: Week 4 (n=32, 31) | 0.4727 (0.43270) | 0.3548 (0.36529)
  Reflux: CFB Week 4 (n=32, 31) | 0.1328 (0.36469) | 0.0202 (0.26437)
  Reflux: Week 8 (n=32, 31) | 0.4660 (0.39881) | 0.4389 (0.46573)
  Reflux: CFB Week 8 (n=32, 31) | 0.1261 (0.36875) | 0.1043 (0.41664)
  Reflux: Week 12 (n=27, 30) | 0.4306 (0.41069) | 0.3417 (0.33142)
  Reflux: CFB Week 12 (n=27, 30) | 0.0880 (0.35494) | 0.0042 (0.26155)
  Reflux: Week 16 (n=25, 28) | 0.3950 (0.37270) | 0.3348 (0.39682)
  Reflux: CFB Week 16 (n=25, 28) | 0.0750 (0.25259) | -0.0045 (0.31820)
  Distention/Bloating: Baseline (n=32, 31) | 0.3984 (0.57100) | 0.5968 (0.58693)
  Distention/Bloating: Week 4 (n=32, 31) | 0.6406 (0.65049) | 0.4919 (0.65346)
  Distention/Bloating: CFB Week 4 (n=32, 31) | 0.2422 (0.41874) | -0.1048 (0.50734)
  Distention/Bloating: Week 8 (n=32,31) | 0.5703 (0.60985) | 0.4247 (0.57188)
  Distention/Bloating: CFB Week 8 (n=32, 31) | 0.1719 (0.47280) | -0.1720 (0.43245)
  Distention/Bloating: Week 12 (n=27, 30) | 0.5370 (0.70610) | 0.4250 (0.56152)
  Distention/Bloating: CFB Week 12 (n=27, 30) | 0.2130 (0.59929) | -0.1833 (0.47766)
  Distention/Bloating: Week 16 (n=25, 28) | 0.4800 (0.61627) | 0.4286 (0.48523)
  Distention/Bloating: CFB Week 16 (n=25, 28) | 0.1200 (0.45139) | -0.1518 (0.45307)
  Diarrhea: Baseline (n=32, 31) | 0.3281 (0.48542) | 0.2742 (0.48026)
  Diarrhea: Week 4 (n=32, 31) | 0.3125 (0.48775) | 0.2258 (0.48026)
  Diarrhea: CFB Week 4 (n=32, 31) | -0.0156 (0.57480) | -0.0484 (0.43503)
  Diarrhea: Week 8 (n=32, 31) | 0.2813 (0.37968) | 0.3226 (0.55600)
  Diarrhea: CFB Week 8 (n=32, 31) | -0.0469 (0.46419) | 0.0484 (0.58245)
  Diarrhea: Week 12 (n=27, 30) | 0.2778 (0.46685) | 0.2000 (0.48423)
  Diarrhea: CFB Week 12 (n=27, 30) | -0.0556 (0.56045) | -0.0667 (0.58329)
  Diarrhea: Week 16 (n=25, 28) | 0.3400 (0.51478) | 0.2500 (0.51819)
  Diarrhea: CFB Week 16 (n=25, 28) | 0.0400 (0.57591) | -0.0179 (0.61587)
  Social Functioning: Baseline (n=32, 31) | 0.1250 (0.28078) | 0.1893 (0.43585)
  Social Functioning: Week 4 (n=32, 31) | 0.1563 (0.26072) | 0.1775 (0.27199)
  Social Functioning: CFB Week 4 (n=32, 31) | 0.0313 (0.25893) | -0.0118 (0.28143)
  Social Functioning: Week 8 (n=32, 31) | 0.1886 (0.31322) | 0.1936 (0.33647)
  Social Functioning: CFB Week 8 (n=32, 31) | 0.0635 (0.29233) | 0.0044 (0.37997)
  Social Functioning: Week 12 (n=27, 30) | 0.1173 (0.23488) | 0.1944 (0.30028)
  Social Functioning: CFB Week 12 (n=27, 30) | 0.0432 (0.25154) | -0.0011 (0.35730)
  Social Functioning: Week 16 (n=25, 28) | 0.0600 (0.13502) | 0.1667 (0.27596)
  Social Functioning: CFB Week 16 (n=25, 28) | 0.0133 (0.16607) | -0.0131 (0.40515)
  Emotional Wellbeing: Baseline (n=32, 31) | 0.0937 (0.26033) | 0.1326 (0.41910)
  Emotional Wellbeing: Week 4 (n=32, 30) | 0.0937 (0.21697) | 0.0778 (0.32516)
  Emotional Wellbeing: CFB Week 4 (n=32, 30) | 0.0000 (0.17831) | -0.0593 (0.14808)
  Emotional Wellbeing: Week 8 (n=32, 31) | 0.1181 (0.33273) | 0.0825 (0.29680)
  Emotional Wellbeing: CFB Week 8 (n=32, 31) | 0.0243 (0.11887) | -0.0502 (0.19846)
  Emotional Wellbeing: Week 12 (n=27, 30) | 0.0493 (0.13182) | 0.0852 (0.30979)
  Emotional Wellbeing: CFB Week 12 (n=27, 30) | 0.0123 (0.12055) | -0.0482 (0.14786)
  Emotional Wellbeing: Week 16 (n=25, 28) | 0.0266 (0.08030) | 0.0833 (0.39959)
  Emotional Wellbeing: CFB Week 16 (n=25, 28) | 0.0000 (0.10627) | -0.0357 (0.12851)
  Fecal Soilage: Baseline (n=32, 31) | 0.0313 (0.17678) | 0.1290 (0.42755)
  Fecal Soilage: Week 4 (n=32, 31) | 0.0313 (0.17678) | 0.1290 (0.42755)
  Fecal Soilage: CFB Week 4 (n=32, 31) | 0.0000 (0.00000) | 0.0000 (0.00000)
  Fecal Soilage: Week 8 (n=32, 31) | 0.0313 (0.17678) | 0.1613 (0.45437)
  Fecal Soilage: CFB Week 8 (n=32, 31) | 0.0000 (0.00000) | 0.0323 (0.17961)
  Fecal Soilage: Week 12 (n=27, 30) | 0.0370 (0.19245) | 0.1333 (0.43417)
  Fecal Soilage: CFB Week 12 (n=27, 30) | 0.0370 (0.19245) | 0.0000 (0.00000)
  Fecal Soilage: Week 16 (n=25, 28) | 0.0400 (0.20000) | 0.1071 (0.41627)
  Fecal Soilage: CFB Week 16 (n=25, 28) | 0.0400 (0.20000) | 0.0000 (0.00000)
  Constipation: Baseline (n=32, 31) | 0.2422 (0.40899) | 0.1694 (0.26130)
  Constipation: Week 4 (n=32, 30) | 0.2656 (0.34159) | 0.1500 (0.29066)
  Constipation: CFB Week 4 (n=32, 30) | 0.0234 (0.42293) | -0.0250 (0.30336)
  Constipation: Week 8 (n=32, 31) | 0.2578 (0.39901) | 0.1613 (0.46345)
  Constipation: CFB Week 8 (n=32, 31) | 0.0156 (0.25350) | -0.0081 (0.38989)
  Constipation: Week 12 (n=27, 30) | 0.2407 (0.38904) | 0.2111 (0.36075)
  Constipation: CFB Week 12 (n=27, 30) | 0.0370 (0.37148) | 0.0528 (0.49008)
  Constipation: Week 16 (n=25, 28) | 0.1800 (0.29333) | 0.1518 (0.27504)
  Constipation: CFB Week 16 (n=25, 28) | 0.0200 (0.37444) | -0.0179 (0.42453)
  Total Score: Baseline (n=32, 31) | 0.2194 (0.24262) | 0.2761 (0.32679)
  Total Score: Week 4 (n=32, 31) | 0.2845 (0.28528) | 0.2432 (0.31264)
  Total Score: CFB Week 4 (n=32, 31) | 0.0651 (0.20058) | -0.0330 (0.13591)
  Total Score: Week 8 (n=32, 31) | 0.2759 (0.26133) | 0.2706 (0.29132)
  Total Score: CFB Week 8 (n=32, 31) | 0.0564 (0.15749) | -0.0055 (0.20053)
  Total Score: Week 12 (n=27, 30) | 0.2416 (0.25329) | 0.2299 (0.27136)
  Total Score: CFB Week 12 (n=27, 30) | 0.0564 (0.16790) | -0.0492 (0.17709)
  Total Score: Week 16 (n=25, 28) | 0.2237 (0.19767) | 0.2284 (0.26906)
  Total Score: CFB Week 16 (n=25, 28) | 0.0481 (0.14444) | -0.0372 (0.20737)

ADVERSE EVENTS:
Time Frame: From baseline up to 28 days after the last dose of study drug (last dose = Week 16)
Arm/Group | Pirfenidone: 2-Week Titration Group | Pirfenidone: 4-Week Titration Group
Serious Adverse Events (participants affected / at risk) | 3/32 | 0/31
Other Adverse Events (participants affected / at risk) | 31/32 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone: 2-Week Titration Group (N=32) | Pirfenidone: 4-Week Titration Group (N=31)
Bronchitis (Infections and infestations) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone: 2-Week Titration Group (N=32) | Pirfenidone: 4-Week Titration Group (N=31)
Palpitations (Cardiac disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 16 | 15
Stomach discomfort (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 9 | 9
Asthenia (General disorders) | 2 | 5
Chest discomfort (General disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 13 | 10
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 3
Weight decreased (Investigations) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 14 | 14
Hypoaesthesia (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 5
Hot flush (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.